CLINICAL TRIAL: NCT06072209
Title: Long-term Effects of an Online Intervention Targeting Depression and Reward Sensitivity - Predictors and Mechanisms of Treatment Success
Brief Title: Long-term Effects ReSet Your Mind - Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: ReSet your Mind - Mechanisms
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Depression Mild; Depression Moderate
Keywords: reward sensitivity; reward processing; depression; randomized controlled trial; online intervention; behavioral activation; mindfulness; gratitude
MeSH Terms: conditions — Depression | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Behavioral Activation (Experimental): 14 days of daily excercises
  Interventions: Behavioral: Behavioral Activation
- Mindfulness and Gratitude (Experimental): 14 days of daily excercises
  Interventions: Behavioral: Mindfulness and Gratitude
- Combination: Behavioral Activation and Mindfulness and Gratitude (Experimental): 14 days of daily excercises
  Interventions: Behavioral: Combination of Behavioral Activation and Mindfulness and Gratitude
- Waitlist control group (No Intervention): Will receive the intervention (combination) after two weeks of intervention time of the other groups.

INTERVENTIONS:
Behavioral: Behavioral Activation — - instruction to create a list of individual positive activities. - instruction to include daily positive activities and fill out a mood protocol, which covers the time period shortly before, during and after the activity.
  Arms: Behavioral Activation
Behavioral: Mindfulness and Gratitude — - instruction to fill out a mindfulness diary: reflection of daily pleasant situation, instructing the participants to revisit the impressions of their 5 senses during this situation, in addition they should specify how long they have actually dealt with
  Arms: Mindfulness and Gratitude
Behavioral: Combination of Behavioral Activation and Mindfulness and Gratitude — This group will do a combination of the two intervention types.
  Arms: Combination: Behavioral Activation and Mindfulness and Gratitude

SUMMARY:
See: ClinicalTrials.gov ID: NCT05402150

Relevant for this Paper:

This investigation aims to evaluate the stability of the effectiveness of different two-week online interventions in a four months follow-up regarding reward sensitivity, anhedonia and depression.

The authors will further investigate factors influencing treatment success regarding reward sensitivity. The investigators assume that the more depressive expectations and stress improve during our online intervention, the more change in reward insensitivity is experienced at follow-up. In addition, it is hypothesized that the more people engaged in physical activities and social encounters during the two-week online intervention, the more change in reward insensitivity is experienced at follow-up.

DETAILED DESCRIPTION:
See for main study: ClinicalTrials.gov ID: NCT05402150.

A possible maintaining role in depressive symptoms plays reward hyposensitivity. Therefore, treatments should include evidence-based psychological interventions that target and modify reward insensitivity. Prior research lacks studies investigating reward sensitivity as main outcome measure, especially in the web-based format. This is why this study investigated an online intervention with the following groups regarding effectively increasing reward sensitivity compared to a waitlist control condition:

a) mindfulness-based interventions, b) behavioral activation, c) a combination of both.

The daily exercises were supported via videos and worksheets. Here, the investigators explore the effects after a four-months follow-up. In addition, this paper will deal with the long-term prediction of reward sensitivity, a feature not considered in our main paper preregistered with the ID NCT05402150. Factors, which are considered to play a big role in reward sensitivity are perceived stress, depressive expectations, physical activity and the frequency of social encounters.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Fluent in German
* Informed consent
* Depressive symptoms (PHQ-9 > 5)

Exclusion Criteria:

* suicidality, severe depression
* current or lifetime: substance use disorder, psychotic disorders, bipolar I or II
* current psychotherapy
* if antidepressant medication: has not been stable over the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms (Patient Health Questionnaire-9, PHQ-9) | baseline, post intervention (after 2 weeks), 4 months follow-up
  * Items range from 0 to 3 (0 = not at all; 1 = several days; 2 = more than a week; 3 = nearly every day).
  * PHQ-9 total score ranges from 0 to 27 (classification of scores: 5-9 mild depression; 10-14 as moderate depression; 15-19: moderately severe depression; 20 - 27 severe depression).
  * Consequently, a higher score means worse depressive symptoms.
Reward sensitivity (Positive Valence System Scale-21, PVSS-21) | baseline, post intervention (after 2 weeks), 4 months follow-up
  * Items range from 1 to 9 (1 = extremely untrue of me, 2 = very untrue of me, 3 = moderately untrue of me, 4 = slightly untrue of me, 5 = neutral, 6 = slightly true of me, 7 = moderately true of me, 8 = very true of me, 9 = extremely true of me).
  * PVSS-21 total score ranges from 21 to 189.
  * Consequently, a higher score means a higher reward responding.
Anhedonia (Snaith-Hamilton-Pleasure-Scale, SHAPS-D) | baseline, post intervention (after 2 weeks), 4 months follow-up
  * Items range from "Definitely Agree", "Agree", "Disagree", and "Strongly Disagree". Either of the "Disagree responses" receive a score of 1 and either of the "Agree responses" receive a score of 0.
  * SHAPS-D total score ranges from 0 to 14.
  * Consequently, a higher score means a greater state anhedonia.
Change in Stress level (Perceived-Stress-Scale 10, PSS-10) | baseline, post intervention (after 2 weeks), 4 months follow-up
  * Items range from 1 to 5 (1= never, 2 = almost never, 3 = sometimes, 4 = fairly often, 5 = very often) Items 4, 5, 7 and 8 are reverse scored for the total score.
  * PH=perceived helplessness subscale; PSE=perceived self-efficacy subscale
  * PH subscale is computed by summing up Items 1, 2, 3, 6, 9 and 10; the PSE subscale is computed by summing up items 4, 5, 7 and 8
  * PSS-10 total score is the sum of all PH and reversed PSE items
  * Consequently, a higher score means a greater level of stress.
Change in Depressive Expectations (Depressive Expectations Scale, DES) | baseline, post intervention (after 2 weeks), 4 months follow-up
  * Items range from 1 to 5 (1 = I disagree , 2 = I partially disagree, 3 = neutral, 4 = I partially agree, 5 = I agree).
  * DES total score ranges from 25 to 125
  * Consequently, a higher score means more dysfunctional depressive expectations.
Amount of physical activity reported during intervention exercises | during intervention
  - Type of activities and reflected pleasant situations that have been selected in the daily online surveys
Amount of social encounters reported during intervention exercises | during intervention
  - Type of activities and reflected pleasant situations that have been selected in the daily online surveys

SECONDARY OUTCOMES:
Personality traits (Big Five Inventory 10, BFI-10) | Baseline, post intervention (after 2 weeks), four months follow-up]
  * Items range from 1 (disagree strongly) to 5 (agree strongly).
  * Scales: openness to experience, conscientiousness, extraversion, agreeableness and neuroticism
Adherence | post intervention (after 2 weeks), 4 months follow-up
  * Number of completed online surveys regarding the intervention exercises (T1 to T14: daily online surveys over the course of two weeks)
  * Self report of implementation of daily exercises in post intervention survey and follow up survey.
Treatment expectation (Generic Rating for Treatment Pre-Experiences, Treatment Expectations, and Treatment Effects, G-EEE) | Baseline, post intervention (after 2 weeks), 4 months follow-up
  - Items range from 0 to 10 (depending on the item from "no improvement" to "greatest improvement imaginable", from "no worsening" to "greatest worsening imaginable", from "no complaints" to "greatest complaints imaginable") and one item, where previous treatment experience is assessed via a choice of "I have never experienced this treatment." (continue with question 8), "I have experienced this treatment during the last 12 months (nearly) daily.", "I have experienced this treatment during the last 12 months on more than 10 days.", "I have experienced this treatment during the last 12 months on about 5 to 10 days.", I have experienced this treatment during the last 12 months on about 1 to 4 days." And "I have not experienced this treatment during the last 12 months, but I have experienced it before."
Treatment credibility and expectancy (Credibility/Expectancy Questionnaire, CEQ) | Baseline
  * Items range from 1 to 9 (Item 1 of Set 1: 1= not at all logical, 5 = somewhat logical, 9 = very logical, Item 2 of Set
    1: 1= not at all useful, 5 = somewhat useful, 9 = very useful, Item 3 of Set 1: 1 = not at all confident, 5 = somewhat confident, 9 = very confident, Item 1 of Set 2: 1 = not at all, 5 = somewhat, 9 = very much), Item 4 of Set 1 and Item 2 of Set 2 give a choice of 0% to 100% in steps of 10 %.
  * CEQ composite score can be derived for each factor (expectancy and credibility)
Trait reward responsiveness (Reward Responsiveness Scale, RRS) | Baseline, post intervention (after 2 weeks), 4 months follow-up
  * Items range from 1 to 4 (1= strong disagreement, 2 = mild disagreement, 3 = mild agreement, 4 = strong agreement)
  * RRS total score ranges from 8 to 32.
  * Consequently, a higher score means a higher reward responsiveness.

OTHER OUTCOMES:
Sociodemographic variables | baseline
  - Gender, age, education, employment, medication, self report lifetime diagnosis of psychiatric conditions, previous experience with psychotherapy etc.
Perceived system usability (System usability Scale, SUS), general feedback about the online intervention | post intervention (after 2 weeks)
  * Items of the SUS range from 1 to 5 (1= strongly disagree to 5 = strongly agree).
  * After a computation, the SUS score can range from 0 to 100. A SUS score above a 68 is considered above average.
  * general feedback about the online intervention: free text entries about the online intervention: criticism, change requests, praise, one closed question: "Would you recommend the online intervention to someone else?" Yes/No
Problems and obstacles during the intervention | post intervention (after 2 weeks)
  - Frequency of telephone contacts made with the principal contact person (Laura Potsch) and specified problems with the implementation of the daily excercises in the daily online survey

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Prof. Dr., Principal Investigator — Dept. of Clinical Psychology and Psychotherapy, Philipps-University Marburg, Germany
Locations (1):
- Philipps University, Marburg, Germany

IPD SHARING:
Plan to Share IPD: No